CLINICAL TRIAL: NCT06235671
Title: The Effects of Upper Cervical Chiropractic Care in Adult Cancer Survivors With Chronic Cancer-related Fatigue: a Feasibility Trial
Brief Title: Effects of Chiropractic on Chronic Cancer-related Fatigue
Acronym: CAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-0029
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Cancer; Fatigue
Keywords: cancer survivors; upper cervical chiropractic; manipulation; cancer-related fatigue; autonomic nervous system
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Intervention Model Description: Single-arm feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chiropractic intervention (Experimental): Upper cervical chiropractic care
  Interventions: Procedure: Chiropractic care

INTERVENTIONS:
Procedure: Chiropractic care — 6 weeks of chiropractic care

SUMMARY:
The primary aims of the proposed trial are centered around examining the feasibility of conducting a prospective, chiropractic intervention study on a population of cancer survivors living in and around Atlanta, Georgia. This includes evaluating various implementation outcomes including recruitment, adherence, tolerability, retention, acceptability, and data fidelity. The results of this trial will inform the design of a future randomized controlled trial (RCT) that has an increased focus on the efficacy/effectiveness of chiropractic care on chronic cancer-related fatigue (CCRF) and other cancer-related sequelae in cancer survivors.

DETAILED DESCRIPTION:
Cancer remission is often marked by the cessation of curative-intent treatments (e.g., surgery, chemotherapy, radiotherapy, immunotherapy), however, troublesome signs and symptoms (e.g., fatigue, depression, cognitive impairment, dysautonomia) related to the cancer and its treatments commonly persist for prolonged periods (i.e., months to years). Of these, chronic cancer-related fatigue (CCRF) is one of the most frequently reported and debilitating symptoms. CCRF may be characterized as tiredness or exhaustion persisting for 3 or more months following the completion of the primary curative-intent cancer therapies which is independent on one's quantity or quality of rest and causes impairments in daily functioning and quality of life. Notably, although the mechanisms underlying CCRF are still unclear, there is some evidence that it may be related to autonomic dysregulation.

Irrespective of the cause(s), lack of identification of and treatment for CCRF and other chronic cancer-related sequelae is commonplace. Further, empirical data supporting the efficacy of interventions to remediate these issues are relatively sparse and urgently needed as the global population of cancer survivors continues to increase. Of note, although there is no universally accepted definition of 'cancer survivor', the investigators define it here as someone who has completed their primary curative-intent therapies and is cancer-free (i.e., has no evidence of active disease). This definition is in line with that of the European Organisation of Research & Treatment of Cancer (EORTC) Survivorship Task Force and the EORTC Quality of Life Group.

Interestingly, a recent study suggested that a single chiropractic adjustment may mitigate lower extremity muscular fatigue during isometric exercise in young, healthy males. However, to the investigators' knowledge, the impact of chiropractic care on CCRF and other health-related challenges that burden cancer survivors has yet to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide written informed consent in English
* 18-65 years of age
* Informed by primary health care provider that there is no evidence of active disease (this is sometimes referred to as "complete remission" or "cured")
* Minimum of 3 months since completion of primary curative-intent cancer therapies including surgery, chemotherapy, radiotherapy, and/or immunotherapy (long-term hormonal therapy permitted)
* Onset of fatigue occurred at some point during illness and/or treatment
* FACIT-Fatigue scale score in the moderate-to-severe range (i.e., at or above the 60th percentile)
* If on any prescription medication (including hormonal therapy), on a stable dose for a minimum of 12 weeks with no plans to change medications or doses during the study

Exclusion Criteria:

* Taking any short-acting benzodiazepine including midazolam & triazolam
* Known disorder resulting in syncope/fainting during postural changes (e.g., postural orthostatic tachycardia syndrome, orthostatic hypotension)
* Pacemaker or known heart condition that influences the electrical or mechanical function of the heart (e.g., severe heart valve disease)
* Diagnosed with an externalizing (e.g., substance use, antisocial disorder) or thought (e.g., schizophrenia, paranoid personality, bipolar) disorder that is uncontrolled or untreated
* Diagnosed with rheumatoid arthritis, osteoporosis, or cervical spine instability
* Currently pregnant
* Current litigation related to a physical, health-related injury
* Chronic pain rated at least 3/10 on a visual analog scale (VAS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment | 6-month data collection period
  Average number of participants recruited/enrolled per month
Participant scheduling | 6-month data collection period
  Average time lag between first lab assessment & first chiropractic visit
Participant compliance | 6-month data collection period
  Proportion of participants violating 1 or more pre-assessment lifestyle restrictions & unable/unwilling to be rescheduled
Participant adherence | 6-month data collection period
  Proportion of participants not attending at least 80% of their chiropractic sessions
Participant tolerability | 6-month data collection period
  Proportion of participants unable/unwilling to complete a given assessment
Participant retention | 6-month data collection period
  Proportion of participants completing the trial
Assessment acceptability | 6-month data collection period
  Most common patient-related acceptability score for each assessment process/procedure
Data fidelity | 6-month data collection period
  Proportion of acquisitions from a given assessment that are unsuitable for analysis
Implementation acceptability | 6-month data collection period
  Most common clinician-rated acceptability score for each trial process/procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yori Gidron, PhD, Principal Investigator — University of Haifa
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No